CLINICAL TRIAL: NCT07344935
Title: Evaluation of the Effectiveness of the Ezisurg Stapling (Ezi Endo Lite) During Laparoscopic Nissen Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ezisurg Medical Co. Ltd. (Other)
Collaborators: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESM-MDR-VIII 1005B
Record Dates: First submitted 2025-12-22; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ezisurg stapler (Experimental): easyEndoTM Lite Linear Cutting Stapler (U12L60) and Loading Units (N60G) manufactured by Ezisurg
  Interventions: Procedure: Ezisurg stapler SLEEVE technique
- Ethicon Stapler (Active Comparator): ECHELON™ Powered Stapler and reload (GST60G) manufactured by Johnson & Johnson.
  Interventions: Procedure: Ethicon Stapler SLEEVE technique

INTERVENTIONS:
Procedure: Ezisurg stapler SLEEVE technique — The Nissen Sleeve technique consists of creating a gastric total fundoplication (Nissen technique) before to perform the removal of 2/3 of the stomach (SLEEVE technique)
  Arms: Ezisurg stapler
Procedure: Ethicon Stapler SLEEVE technique — The Nissen Sleeve technique consists of creating a gastric total fundoplication (Nissen technique) before to perform the removal of 2/3 of the stomach (SLEEVE technique)
  Arms: Ethicon Stapler

SUMMARY:
The Nissen Sleeve technique consists of creating a gastric total fundoplication (Nissen technique) before to perform the removal of 2/3 of the stomach (SLEEVE technique), intends for decrease the rate of gastroesophageal reflux disease (GERD). This study aims to evaluate the influence of the Nissen Sleeve technique on GERD. However, the Ezisurg easyEndoTM Linear Cutting Stapler and Loading Units for Single Use were used in this study, and its safety and performance could be evaluated at the same time.

ELIGIBILITY:
Inclusion Criteria

* Body Mass Index (BMI) ≥ 30 kg/m² (or BMI ≥ 27 kg/m² with at least one obesity-related comorbidity, e.g., type 2 diabetes, hypertension, dyslipidemia).
* Medically eligible for laparoscopic sleeve gastrectomy (LSG) or Nissan sleeve surgery, as determined by a multidisciplinary bariatric team (e.g., surgeon, endocrinologist, dietitian).
* Ability to understand and voluntarily sign written informed consent.
* Willingness to comply with post-operative follow-up protocols (e.g., dietary monitoring, clinical visits, laboratory tests).

Exclusion Criteria

* BMI < 30 kg/m² (or < 27 kg/m² without obesity-related comorbidities).
* Contraindications to laparoscopic surgery (e.g., severe abdominal adhesions, hemodynamic instability, uncorrected coagulopathy).
* History of major gastrointestinal surgery (e.g., gastric bypass, colectomy) or anatomical abnormalities precluding sleeve gastrectomy.
* Active or uncontrolled chronic diseases (e.g., end-stage renal disease, cirrhosis, metastatic cancer, severe cardiovascular disease).
* Psychiatric disorders limiting adherence to post-operative care (e.g., severe depression, psychosis, substance use disorder).
* Pregnancy or breastfeeding (or plans for pregnancy within 12 months post-surgery).
* Allergy or intolerance to surgical materials, anesthesia, or post-operative medications required for the study.
* Inability to communicate or cooperate with study procedures (e.g., language barriers, cognitive impairment).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
The rate of patients with GERD at 24 months | 24 months
  The main objective of the study was to evaluate the impact of Sleeve Gastrectomy procedure with a Nissen fundoplication (Nissen-Sleeve) on the rate of patients with GERD at 24 months.

SECONDARY OUTCOMES:
Surgery time | Perioperative/Periprocedural
Intra-operation incidents | Perioperative/Periprocedural
Hospital stays | Perioperative/Periprocedural
Rate of re-intervention | two-year
Rate of re-hospital | two-year
One-year Endoscopy finding | One-year
Early & Long term post-operative complication | two-year

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Français du Levant, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No